CLINICAL TRIAL: NCT01925989
Title: Evaluation of the Effects of Insulin Peglispro (LY2605541) on Respiratory Quotient During Sleep and Response to Hyperinsulinemia Compared With That of Insulin Glargine in Patients With Type 1 Diabetes Mellitus
Brief Title: A Study of How Insulin Peglispro (LY2605541) and Insulin Glargine Affect the Breakdown of Fat and Sugar in Type 1 Diabetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 14872; I2R-MC-BIDO (Other: Eli Lilly and Company); NCT02211586 (obsolete NCT alias)
Record Dates: First submitted 2013-08-16; First posted 2013-08-20 (Estimated); Results first posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2018-10

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — LY2605541; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Insulin Peglispro/Insulin Glargine (Experimental): Insulin peglispro (LY2605541) administered to participants with T1DM subcutaneously (SQ) once daily (QD) for 28 to 35 days in one of two treatment periods. Dose is based on participant's prestudy basal insulin dosing regimen. Insulin glargine administered to participants with T1DM SQ QD for 28 to 35 days in one of two treatment periods. Dose is based on participant's prestudy basal insulin dosing regimen. Participants continue to use mealtime insulin.
  Interventions: Biological: LY2605541
- Insulin Glargine/Insulin Peglispro (Active Comparator): Insulin glargine administered to participants with T1DM SQ QD for 28 to 35 days in one of two treatment periods. Dose is based on participant's prestudy basal insulin dosing regimen. Participants continue to use mealtime insulin. Insulin peglispro (LY2605541) administered to participants with T1DM subcutaneously (SQ) once daily (QD) for 28 to 35 days in one of two treatment periods. Dose is based on participant's prestudy basal insulin dosing regimen.
  Interventions: Biological: Insulin Glargine
- Control (No Intervention): Control Arm. Untreated healthy participants.

INTERVENTIONS:
Biological: LY2605541 — Administered SQ
  Arms: Insulin Peglispro/Insulin Glargine
Biological: Insulin Glargine — Administered SQ
  Arms: Insulin Glargine/Insulin Peglispro

SUMMARY:
This is a two-period study of participants with type 1 diabetes mellitus (T1DM). In each period, participants will receive once daily injections of stable dose LY2605541 or insulin glargine for 28 to 35 days followed by procedures to look at how the body uses or stores fats and sugars. Participants will continue to use meal time insulin throughout the study. Healthy participants will also enroll in the study. They will not receive any study medication.

ELIGIBILITY:
Inclusion Criteria:

Type 1 Diabetics:

- T1DM for more than 1 year with Hemoglobin A1c (HbA1c) of less than 9.5%

All Participants:

* Otherwise fit and healthy
* Non smoker

Exclusion Criteria:

Type 1 Diabetics:

* Taking medication or supplements other than insulin to control diabetes
* Suffered a hypoglycemic event in the last 12 months that required hospitalization or have poor awareness of hypoglycemia

All Participants:

- Taking fibrates, thyroid replacement therapy, testosterone, beta blockers or systemic corticosteroids

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2013-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence Insulin Peglispro/Insulin Glargine: Insulin peglispro (LY2605541) administered to participants with T1DM subcutaneously (SQ) once daily (QD) for 28 to 35 days in one of two treatment periods. Dose based on participant's prestudy basal insulin dosing regimen. Insulin glargine administered to participants with T1DM SQ QD for 28 to 35 days in one of two treatment periods. Dose based on participant's prestudy basal insulin dosing regimen. Participants continue to use mealtime insulin.
- Sequence Insulin Glargine/Insulin Peglispro: Insulin glargine administered to participants with T1DM SQ QD for 28 to 35 days in one of two treatment periods. Dose based on participant's prestudy basal insulin dosing regimen. Participants continue to use mealtime insulin.Insulin peglispro (LY2605541) administered to participants with T1DM subcutaneously (SQ) once daily (QD) for 28 to 35 days in one of two treatment periods. Dose based on participant's prestudy basal insulin dosing regimen.
- Control: Untreated healthy participants who received no study drug.
Period: Period 1
Arm/Group | Sequence Insulin Peglispro/Insulin Glargine | Sequence Insulin Glargine/Insulin Peglispro | Control
Started | 7 | 8 | 12
Received at Least 1 Dose of Study Drug | 7 | 8 | 0
Completed | 6 | 6 | 12
Not Completed | 1 | 2 | 0
Not completed — Sponsor Decision | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Period: Period 2
Arm/Group | Sequence Insulin Peglispro/Insulin Glargine | Sequence Insulin Glargine/Insulin Peglispro | Control
Started | 6 | 6 | 12
Completed | 6 | 6 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All T1DM: Participants with T1DM who received Insulin peglispro (LY260551) and insulin glargine SQ in either sequence group.
- Total: Total of all reporting groups
Arm/Group | All T1DM | Control | Total
Number analyzed (Participants) | 15 | 12 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (12.2) | 36.9 (12.4) | 36.7 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 8 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 11 | 9 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 14 | 8 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 12 | 27

OUTCOME MEASURES:

1. Primary Outcome: Sleep Respiratory Quotient (RQ) in Type 1 Diabetes Mellitus (T1DM)
Description: Lipid or glucose metabolism was assessed by the measurement of respiratory quotient (RQ) during sleep using whole room calorimetry. RQ is a calculation of basal metabolic rate (BMR) when estimated from carbon dioxide production. It is calculated from the ratio of carbon dioxide produced by the body to oxygen consumed by the body using whole room calorimetry (WRC).
Time Frame: Day 30 post dose, overnight period (0000 to 0600 hours)
Population: All randomized participants with T1DM that received at least 1 dose of study drug. Data from 2 participants could not be used: one due to uncontrolled blood glucose and one due to an increase in thyroid medication.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Insulin Peglispro: Insulin peglispro (LY2605541) administered to participants with T1DM subcutaneously (SQ) once daily (QD) for 28 to 35 days in one of two treatment periods. Dose based on participant's prestudy basal insulin dosing regimen.
- Insulin Glargine: Insulin glargine administered to participants with T1DM SQ QD for 28 to 35 days in one of two treatment periods. Dose based on participant's prestudy basal insulin dosing regimen.
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 13 | 12
ratio | 0.822 (0.026) | 0.846 (0.033)

2. Secondary Outcome: Lipid Oxidation in T1DM and Healthy Participants
Description: Lipid oxidation is derived from RQ, basal metabolic rate and urinary nitrogen, a value of 0.7 indicates that lipids are being metabolized.
Time Frame: Day 30 post dose, overnight period (0000 to 0600 hours)
Population: All randomized participants.
Measure: Mean (Standard Deviation); unit: grams per day (g/day)
Arm/Group | Insulin Peglispro | Insulin Glargine | Control
Number analyzed (Participants) | 13 | 12 | 12
grams per day (g/day) | 0.892 (0.024) | 0.900 (0.024) | 0.906 (0.020)

3. Secondary Outcome: Basal Metabolic Rate (BMR) for T1DM
Description: BMR is the metabolic rate determined at rest 12 to 14 hours after the last meal.
Time Frame: Day 30 post dose, overnight period (0000 to 0600 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 13 | 12
kcal/day | 1511.0 (228.3) | 1403.6 (207.7)

4. Secondary Outcome: Sleep Respiratory Quotient (RQ) of Untreated Healthy Participants
Description: The respiratory quotient (or RQ or respiratory coefficient), is a number used in calculations of basal metabolic rate (BMR) when estimated from carbon dioxide production. It is calculated from the ratio of carbon dioxide produced by the body to oxygen consumed by the body using whole room calorimetry. The overnight period was averaged based on all 1-minutes interval measurements for the duration of the overnight period.
Time Frame: Day 5, overnight period (0000 to 0600 hours)
Population: All randomized, health participant who received no study drug.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Control
Number analyzed (Participants) | 12
ratio | 0.848 (0.020)

5. Secondary Outcome: Total Number of Minutes of Lipid Oxidation (RQ Below 7.6) in T1DM and Healthy Participants
Description: The respiratory quotient (or RQ or respiratory coefficient), is a number used in calculations of basal metabolic rate (BMR) when estimated from carbon dioxide production. It is calculated from the ratio of carbon dioxide produced by the body to oxygen consumed by the body using whole room calorimetry.It is calculated from the ratio of carbon dioxide produced by the body to oxygen consumed by the body using whole data based on all 1-minutes interval measurements for the duration of the overnight period.
Time Frame: Day 5, every minute through 23 hour period
Population: All randomized participants: T1DM participants that received at least 1 dose of study drug, Data from 2 participants could not be used:one due to uncontrolled blood glucose and one due to an increase in thyroid medication,data from 2 participants could not be used: 1 due to uncontrolled blood glucose and 1 due to an increase in thyroid medication.
Measure: Median (Full Range); unit: minutes
Groups:
- Insulin Glargine/Insulin Peglispro: Insulin glargine administered to participants with T1DM SQ QD for 28 to 35 days in one of two treatment periods. Dose is based on participant's prestudy basal insulin dosing regimen.
Arm/Group | Insulin Peglispro | Insulin Glargine/Insulin Peglispro | Control
Number analyzed (Participants) | 13 | 12 | 12
minutes | 22 [3 to 205] | 8 [0 to 61] | 4.5 [0 to 84]

6. Secondary Outcome: Change in RQ, Pre-breakfast to Post-breakfast Meal, in T1DM
Description: The respiratory quotient (or RQ or respiratory coefficient), is a number used in calculations of basal metabolic rate (BMR) when estimated from carbon dioxide production. It is calculated from the ratio of carbon dioxide produced by the body to oxygen consumed by the body using whole room calorimetry.
Time Frame: Day 30 0830 to 0854 hours, Day 30 1000 to 1054 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Insulin Peglispro: Insulin peglispro (LY2605541) administered to participants with T1DM subcutaneously (SQ) once daily (QD) for 28 to 35 days in one of two treatment periods. Dose is based on participant's prestudy basal insulin dosing regimen.
- Insulin Glargine: Insulin glargine administered to participants with T1DM SQ QD for 28 to 35 days in one of two treatment periods. Dose is based on participant's prestudy basal insulin dosing regimen.
Arm/Group | Insulin Peglispro | Insulin Glargine
Number analyzed (Participants) | 11 | 12
ratio | 0.836 (0.055) | 0.874 (0.033)

ADVERSE EVENTS:
Description: One participant in the Insulin Glargine/Insulin Peglispro arm withdrew consent prior to being dosed with study drug and is included in the AE section.
Groups:
- Insulin Peglispro: Insulin peglispro (LY2605541) administered to participants with T1DM subcutaneously (SQ) once daily (QD) for 28 to 35 days in one of two treatment periods. Dose is based on participant's prestudy basal insulin dosing regimen. Participants continue to use mealtime insulin.
- Insulin Glargine: Insulin glargine administered to participants with T1DM SQ QD for 28 to 35 days in one of two treatment periods. Dose is based on participant's prestudy basal insulin dosing regimen. Participants continue to use mealtime insulin.
Arm/Group | Insulin Peglispro | Insulin Glargine | Control
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15 | 0/12
Other Adverse Events (participants affected / at risk) | 5/13 | 3/15 | 1/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Peglispro (N=13) | Insulin Glargine (N=15) | Control (N=12)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 3 (3) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
One participant in the Insulin Glargine/Insulin Peglispro arm withdrew consent prior to being dosed with study drug and is included in the Adverse Event (AE) section.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days